CLINICAL TRIAL: NCT01067742
Title: The Natural History of Mucolipidosis Type IV
Status: Terminated | Type: Observational
Why Stopped: PI left site
Sponsor: Baylor Research Institute (Other)
Collaborators: Rare Diseases Clinical Research Network (Network); National Center for Advancing Translational Sciences (NCATS) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 008-295; U54NS065768 (NIH)
Record Dates: First submitted 2010-02-10; First posted 2010-02-12 (Estimated); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Mucolipidosis Type IV
Keywords: Mucolipidosis, retinal dystrophy, mucolipin-1,; lysosomal storage disease, gastrin, mental retardation,; dysmyelination, dysplastic corpus callosum,corneal clouding
MeSH Terms: conditions — Mucolipidoses; Retinal Dystrophies; Lysosomal Storage Diseases; Intellectual Disability; Demyelinating Diseases; Agenesis of Corpus Callosum; Corneal Opacity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, urine and skin
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects with Mucolipidosis Type IV

SUMMARY:
The purpose of this study is to define the natural history of Mucolipidosis Type IV and identify potential clinical outcome measures.

DETAILED DESCRIPTION:
Mucolipidosis type IV (MLIV) is an autosomal recessive disorder typically characterized by severe psychomotor delay evident by the end of the first year of life and slowly progressive visual impairment during the first decade as a result of a combination of corneal clouding and retinal degeneration. By the end of the first decade of life, and always by their early teens, individuals with typical MLIV develop severe visual impairment as a result of retinal degeneration. MLIV is an under-diagnosed and unique lysosomal disorder in that it often is mistaken either for cerebral palsy or for a retinal dystrophy of unknown cause. In addition, it is caused by a defect in a cation channel rather than by a lysosomal hydrolase. This study represents the only prospective clinical study in this patient population. Now that an animal model has been created and novel therapies will likely be tested, it is particularly important to define the natural history of this disorder and identify potential clinical outcome measures.

ELIGIBILITY:
Inclusion Criteria:

Subjects must:

* Have a definitive diagnosis of MLIV based at least on a compatible history and significantly elevated blood gastrin levels
* Be able to travel to the Baylor Institute of Metabolic Disease in Dallas and spend 2-3 working days on site
* Be able to tolerate a general exam and neurological exam
* Be able to tolerate a modest amount of blood drawing, provide a urine specimen, and have a skin biopsy(if not previously done)
* Be able to tolerate the performance of necessary neuroimaging studies to include EEG and Head MRI
* Be able to tolerate a neuropsychological testing and rehabilitation evaluation

Exclusion Criteria:

-

Ages: 1 Year to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects previously identified with Mucolipidosis Type IV
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2009-02-19 (Actual); Primary Completion 2021-07-07 (Actual); Study Completion 2021-07-07 (Actual)

PRIMARY OUTCOMES:
Neuropsychological testing | Annual by 5 years

SECONDARY OUTCOMES:
Blood tests | Annual by 5 years
Urine tests | Annual by 5 years
MRI of the brain | Annual by 5 years
Rehabilitation evaluation | Annual by 5 years
Nutritional status evaluation | Annual by 5 years
Skin biopsy | 1 year only

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor Institute of Metabolic Disease, Dallas, Texas, United States

REFERENCES:
- [Derived] Cougnoux A, Drummond RA, Fellmeth M, Navid F, Collar AL, Iben J, Kulkarni AB, Pickel J, Schiffmann R, Wassif CA, Cawley NX, Lionakis MS, Porter FD. Unique molecular signature in mucolipidosis type IV microglia. J Neuroinflammation. 2019 Dec 28;16(1):276. doi: 10.1186/s12974-019-1672-4. PMID 31883529